CLINICAL TRIAL: NCT07374874
Title: A Cohort Study on the Association Between the Autonomic Nervous System Function and Acute GvHD After Patients Receiving Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: A Cohort Study on the Association Between the ANS Function and Acute GvHD
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: IIT2025112
Record Dates: First submitted 2025-11-28; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Transplant-Related Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients receiving HLA-haploidentical transplants

SUMMARY:
This is a prospective observational study. The investigators plan to utilize this model as a tool for early classification and interrogate ANS function of transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be > 16 years of age;
2. Patients receiving HLA-haploidentical transplants;
3. Patients have to sign an informed consent form before the start of the research procedure.

Exclusion Criteria:

1. Tandem transplantation or multiple transplantations;
2. Mental or other medical conditions that make the patients unable to comply with the research treatment and monitoring requirements;
3. Patients who are ineligible for the study due to other factors, or will bear great risk if participating in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients receiving HLA-haploidentical transplants at the Institute of Hematology, Chinese Academy of Medical Sciences (IHCAMS)
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Result of heart rate response to standing test | Within one month before the transplantation and during 17-25 days after the transplantation.
  Autonomic nervous system functional tests including heart rate response to standing will be performed within one month before the transplantation and during 17-25 days after the transplantation.
Result of piloerection test | Within one month before the transplantation and during 17-25 days after the transplantation.
  Autonomic nervous system functional tests including piloerection will be performed within one month before the transplantation and during 17-25 days after the transplantation.
Number of participants with abnormal dynamic electrocardiography readings | Within one month before the transplantation and during 17-25 days after the transplantation.
  Dynamic electrocardiography will be performed within one month before the transplantation and during 17-25 days after the transplantation.

SECONDARY OUTCOMES:
Incidence of severe acute GvHD after transplantation within 100 days and incidences of acute GvHD (any grade) in various target organs. | 100 days after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

DOCUMENTS (1):
  • Study Protocol (2025-11-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT07374874/Prot_000.pdf